CLINICAL TRIAL: NCT04466605
Title: Effect of Tele-Yoga Therapy on Patients With Chronic Musculoskeletal Pain During Covid-19 Lockdown: Randomized Clinical Trial
Brief Title: Effect of Tele-Yoga Therapy on Patients With Chronic Musculoskeletal Pain During Covid-19 Lockdown
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: NMP Medical Research Institute (Other); Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AU/NMP/0921
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Tele-Yoga Therapy; Chronic musculoskeletal pain; Randomized controlled trial
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Yoga Therapy (Experimental): All patients randomized to the intervention group had one to one yoga sessions with yoga therapist twice a week for 45 minutes on secure virtual platform. Patients were encouraged with home practice to follow everyday at least for 30-mins.
  Interventions: Other: Tele-yoga therapy
- Usual Care (Active Comparator): Patients randomized to usual care continued to receive care for their chronic musculoskeletal pain from their primary care physician. There was no attempt by to influence clinical management unless an emergency arose
  Interventions: Other: Primary care

INTERVENTIONS:
Other: Tele-yoga therapy — Each session included combinations of different yoga exercises, postures, yoga breathing, yoga relaxation techniques, yoga counselling and meditative practices based on individualisation.
  Arms: Tele-Yoga Therapy
Other: Primary care — Patients will follow standard care provided by primary care physicians including analgesics and self care management.
  Arms: Usual Care

SUMMARY:
Covid-19 outbreak and lockdown measures raised significant concerns over clinical management of chronic pain patients around the world. Patients with chronic musculoskeletal pain (CMSP) are at high risk of physical disability, psychological distress, and poor quality of life. Analgesic medications were main management during lockdown, but opioid-related concerns have prompted to find immediate alternatives.

Present study was undertaken to determine whether patients randomized to tele-yoga therapy would experience less pain, disability and improved global health, adherence and satisfaction, compared with patients assigned to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients having pain that was musculoskeletal, defined as regional (joints, limbs, back, neck) or more generalized (fibromyalgia or chronic widespread pain);
* Persistent pain ( ≥3 months) despite trying conventional treatment.
* Access to virtual platform with internet.
* Ready to give informed consent

Exclusion Criteria:

* Schizophrenia,
* Psychiatric disorder
* Cognitive impairment
* Suicidal ideation
* Current illicit drug use
* Terminal illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Severity of pain | From baseline to 6-week post intervention
  Pain was assessed using the Brief Pain Inventory (BPI), which rates the severity of pain on 4 items (current, worst, least, and average pain in past week)
Interference of pain | From baseline to 6-week post intervention
  Interference of pain in 7 areas (mood, physical activity, work, social activity, relations with others, sleep, enjoyment of life) were reported using BPI

SECONDARY OUTCOMES:
Global rating of change in pain | From baseline to 6-week post interventiona
  7-point global rating of pain change was used to assess change in pain
Intervention specific satisfaction | From baseline to 6-week post interventiona
  10 point scale was used to assess intervention-specific satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Meghwal, Principal Investigator — NMP Medical Research Institute, India; Neha Sharma, Study Director — Aarogyam UK; Bhavna Pandya, Study Chair — Aarogyam UK; Abhimanyu Kumar, Study Chair — Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University
Locations (1):
- NMP Medical Research Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided